CLINICAL TRIAL: NCT03608839
Title: Effect of Dexamethasone on Reduction of Macular Thickness in Diabetic Patients, a Randomized Clinical Trial
Acronym: EDRMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Rodrigo Pessoa Cavalcanti Lira, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2018-07-12; First posted 2018-08-01 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema; Intravitreal dexamethasone solution; Short term treament

STUDY DESIGN:
Intervention Model Description: At the baseline study visit, patients were randomized with a 1:1:1 allocation to receive dexamethasone solution 4 mg/ml: 0,01 ml (40 µg); or 0,03 ml (120 µg); or 0,05 ml (200 µg). In follow up visits (1, 3, 7, 14, 21, 28 days after) were performed BCVA, slit-lamp biomicroscopy, applanation tonometry, fundus biomicroscopy, SD- OCT (Spectralis; Heidelberg Engineering, Heidelberg, Germany). The randomization schedule was computer generated and stored in a locked cabinet until the study ended. Both patients and the study personnel who collected BCVA, OCT data were masked to the patient study assignment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All the patients were masked. They didn't have acess to the group they belonged.
  The care provider didn't know the quantity of the drug injected. The outcome assessor was masked as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0,01ml dexamethasone solution (Experimental): One intravitreous injection of 0,01 ml dexamethasone solution 4 mg/ml.
  Interventions: Drug: Intravitreous Dexamethasone Solution 4mg/ml - vol 0,01 ml
- 0,03 ml dexamethasone solution (Experimental): One intravitreous injection of 0,03 ml dexamethasone solution 4 mg/ml.
  Interventions: Drug: Intravitreous Dexamethasone Solution 4mg/ml - vol 0,03 ml
- 0,05 ml dexamethasone solution (Experimental): One intravitreous injection of 0,05 ml dexamethasone solution 4 mg/ml.
  Interventions: Drug: Intravitreous Dexamethasone Solution 4mg/ml - vol 0,05 ml

INTERVENTIONS:
Drug: Intravitreous Dexamethasone Solution 4mg/ml - vol 0,01 ml — 0,01 ml intravitreous dexamethasone solution 4mg/ml injection.
  Other Names: 0,01 ml intravitreous dexamethasone solution
  Arms: 0,01ml dexamethasone solution
Drug: Intravitreous Dexamethasone Solution 4mg/ml - vol 0,03 ml — 0,03 ml intravitreous dexamethasone solution 4mg/ml injection.
  Other Names: 0,03 ml intravitreous dexamethasone solution
  Arms: 0,03 ml dexamethasone solution
Drug: Intravitreous Dexamethasone Solution 4mg/ml - vol 0,05 ml — 0,05 ml intravitreous dexamethasone solution 4mg/ml injection.
  Other Names: 0,05 ml intravitreous dexamethasone solution
  Arms: 0,05 ml dexamethasone solution

SUMMARY:
Purpose: To determine the impact of short-term 4mg/ml dexamethasone solution treatment in diabetic macular edema (DME).

Design: Phase II, randomized, prospective, parallel, interventional study.

Participants: Pseudophakic patients with central-involved DME.

Methods: Twenty-seven patients with visual impairment caused by DME were randomized in a 1:1:1 ratio, in order to investigate treatment with 0.01 ml, 0.03 ml and 0.05 ml intravitreous dexamethasone solutions, and followed-up over 28 days

Outcome Measures: The primary outcome was macular thickness at three days after intravitreous dexamethasone. The secondary outcomes were macular thickness at 28 days after intravitreous dexamethasone, best-corrected visual acuity (BCVA) and intraocular pressure (IOP) at three and 28 days after intravitreous dexamethasone

DETAILED DESCRIPTION:
This is a prospective, phase II, randomized, interventional, monocentric study. Data of consecutive patients with DME who volunteered to participate in the research at the department of ophthalmology of State University of Campinas (UNICAMP) - Brazil between May 2016 and December 2017 were analysed.

At the screening visit, all patients underwent complete ophthalmic evaluation, including best corrected visual acuity (BCVA), slit-lamp biomicroscopy, applanation tonometry, fundus biomicroscopy, fluorescein angiography (Visucam NM/ FA Carl Zeiss; Carl Zeiss Meditec, California, USA), SD- OCT (Spectralis; Heidelberg Engineering, Heidelberg, Germany). Central macular thickness was obtained through 7 horizontal lines ( 30° x 5° area), centered on the fovea, with 1536 A scans per line at 240 µm intervals.

At the baseline study visit, patients were randomized with a 1:1:1 allocation to receive dexamethasone solution 4 mg/ml: 0,01 ml (40 µg) ; or 0,03 ml (120 µg); or 0,05 ml (200 µg). In follow up visits (1, 3, 7, 14, 21, 28 days after) were performed BCVA, slit-lamp biomicroscopy, applanation tonometry, fundus biomicroscopy, SD- OCT.

ELIGIBILITY:
Inclusion Criteria:

* age > = 18 years;
* diagnosis of DM type 2;
* pseudophakic patients
* presence of clinically significant DME according to ETDRS guidelines;
* best correct visual acuity (BCVA) between 20/400 and 20/40;
* central macular thickness (CMT) >= 300 µm measured by spectral domain optical coherence tomography ( Spectralis® Heidelberg). If both eyes of the patient met the elegibility criteria, the eye with worse BCVA at baseline was designated as the study eye.

Exclusion Criteria:

* any treatment of DME in the previous 4 months;
* pan retinal photocoagulation (PRP) in the previous 4 months or antecipated need of PRP for the next 6 months;
* any ophthalmologic surgery performed in the previous 4 months;
* history of pars plana vitrectomy;
* history of open-angle glaucoma or intraocular pressure elevation induced by corticosteroids that required anti-glaucomatous treatment or anti- hypertensive ocular treatment;
* intraocular pressure >= 21 mmHg;
* patients with characteristics that meet the inclusion criteria, but refused to sign the written general consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo PC Lira, MD, Study Chair — University of Campinas, Brazil
Locations (1):
- State University of Campinas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maturi RK, Glassman AR, Liu D, Beck RW, Bhavsar AR, Bressler NM, Jampol LM, Melia M, Punjabi OS, Salehi-Had H, Sun JK; Diabetic Retinopathy Clinical Research Network. Effect of Adding Dexamethasone to Continued Ranibizumab Treatment in Patients With Persistent Diabetic Macular Edema: A DRCR Network Phase 2 Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jan 1;136(1):29-38. doi: 10.1001/jamaophthalmol.2017.4914. PMID 29127949
- [Background] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Background] Elman MJ, Bressler NM, Qin H, Beck RW, Ferris FL 3rd, Friedman SM, Glassman AR, Scott IU, Stockdale CR, Sun JK; Diabetic Retinopathy Clinical Research Network. Expanded 2-year follow-up of ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):609-14. doi: 10.1016/j.ophtha.2010.12.033. PMID 21459214
- [Background] Tamura H, Miyamoto K, Kiryu J, Miyahara S, Katsuta H, Hirose F, Musashi K, Yoshimura N. Intravitreal injection of corticosteroid attenuates leukostasis and vascular leakage in experimental diabetic retina. Invest Ophthalmol Vis Sci. 2005 Apr;46(4):1440-4. doi: 10.1167/iovs.04-0905. PMID 15790913
- [Background] Wang K, Wang Y, Gao L, Li X, Li M, Guo J. Dexamethasone inhibits leukocyte accumulation and vascular permeability in retina of streptozotocin-induced diabetic rats via reducing vascular endothelial growth factor and intercellular adhesion molecule-1 expression. Biol Pharm Bull. 2008 Aug;31(8):1541-6. doi: 10.1248/bpb.31.1541. PMID 18670086
- [Background] Mitchell P, Bandello F, Schmidt-Erfurth U, Lang GE, Massin P, Schlingemann RO, Sutter F, Simader C, Burian G, Gerstner O, Weichselberger A; RESTORE study group. The RESTORE study: ranibizumab monotherapy or combined with laser versus laser monotherapy for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):615-25. doi: 10.1016/j.ophtha.2011.01.031. PMID 21459215
- [Background] Nguyen QD, Brown DM, Marcus DM, Boyer DS, Patel S, Feiner L, Gibson A, Sy J, Rundle AC, Hopkins JJ, Rubio RG, Ehrlich JS; RISE and RIDE Research Group. Ranibizumab for diabetic macular edema: results from 2 phase III randomized trials: RISE and RIDE. Ophthalmology. 2012 Apr;119(4):789-801. doi: 10.1016/j.ophtha.2011.12.039. Epub 2012 Feb 11. PMID 22330964
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] Bandello F, Battaglia Parodi M, Lanzetta P, Loewenstein A, Massin P, Menchini F, Veritti D. Diabetic macular edema. Dev Ophthalmol. 2010;47:73-110. doi: 10.1159/000320075. Epub 2010 Aug 10. PMID 20703045
- [Background] Kempen JH, O'Colmain BJ, Leske MC, Haffner SM, Klein R, Moss SE, Taylor HR, Hamman RF; Eye Diseases Prevalence Research Group. The prevalence of diabetic retinopathy among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):552-63. doi: 10.1001/archopht.122.4.552. PMID 15078674
- [Derived] Fonseca ALA, Panetta H, Nascimento MA, Lira RPC, Arieta CEL. Effect of intravitreal dexamethasone solution on the reduction of macular thickness in pseudophakic diabetic patients in a public hospital in Brazil: a randomized clinical trial. Clin Ophthalmol. 2019 Aug 9;13:1523-1531. doi: 10.2147/OPTH.S214329. eCollection 2019. PMID 31496644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from DME diagnosed volunteers was collected and analyzed at the Department of Ophthalmology, State University of Campinas (UNICAMP), Brazil between May 2016 and December 2017
Pre-assignment Details: Informed written consent was obtained from all patients, and approved by the ethics committee of the Clinical Hospital of the State University of Campinas
Period: Overall Study
Arm/Group | 0,01ml Dexamethasone Solution | 0,03 ml Dexamethasone Solution | 0,05 ml Dexamethasone Solution
Started | 9 | 9 | 9
Completed | 9 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0,01ml Dexamethasone Solution | 0,03 ml Dexamethasone Solution | 0,05 ml Dexamethasone Solution | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (5.63) | 65.5 (8.26) | 71.3 (7.36) | 67.9 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 12
  Male | 6 | 5 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 9 | 9 | 9 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 9 | 9 | 9 | 27
Eye (Right) [Count of Participants; unit: Participants] | 3 | 7 | 5 | 15
Epirretinal membrane [Count of Participants; unit: Participants] | 5 | 3 | 2 | 10
Subretinal fluid [Count of Participants; unit: Participants] | 1 | 2 | 1 | 4
Microaneurysms in foveal region [Count of Participants; unit: Participants] | 8 | 8 | 9 | 25
Posterior vitreous detachment [Count of Participants; unit: Participants] | 2 | 2 | 5 | 9
Central macular thickness [Mean (Standard Deviation); unit: µm] | 527.6 (154.21) | 630 (254.68) | 453.3 (140.39) | 537.4 (196.94)
Best corrected visual acuity [Mean (Standard Deviation); unit: ETDRS Letters] | 52.5 (13.98) | 47.2 (19.31) | 60 (15.31) | 53.2 (16.61)
Intraocular pressure [Mean (Standard Deviation); unit: mmHg] | 11.8 (2.02) | 13.22 (2.53) | 11.6 (2.55) | 12.2 (2.39)

OUTCOME MEASURES:

1. Primary Outcome: Macular Thickness at 3 Days After Intravitreous Dexamethasone
Description: Measure macular thickness at 3 days after intravitreous dexamethasone with OCT - unit µm
Time Frame: Three days after intravitreous dexamethasone
Population: Macular thickness at 3 days after intravitreous dexamethasone
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | 0,01ml Dexamethasone Solution | 0,03 ml Dexamethasone Solution | 0,05 ml Dexamethasone Solution
Number analyzed (Participants) | 9 | 9 | 9
µm | 438.44 (124.55) | 465.22 (115.25) | 368.22 (126.92)

2. Secondary Outcome: Macular Thickness at 28 Days After Intravitreous Dexamethasone
Description: Measure macular thickness at 28 days after intravitreous dexamethasone with OCT - unit µm
Time Frame: 28 days after intravitreous dexamethasone
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | 0,01ml Dexamethasone Solution | 0,03 ml Dexamethasone Solution | 0,05 ml Dexamethasone Solution
Number analyzed (Participants) | 9 | 9 | 9
µm | 554.66 (175.91) | 617.22 (245.83) | 451.44 (154.48)

3. Secondary Outcome: Best Corrected Visual Acuity (BCVA) at 3 Days After Intravitreous Dexamethasone
Description: Measure best corrected visual acuity (BCVA) at 3 days after intravitreous dexamethasone with ETDRS chart
Time Frame: Three days after intravitreous dexamethasone
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | 0,01ml Dexamethasone Solution | 0,03 ml Dexamethasone Solution | 0,05 ml Dexamethasone Solution
Number analyzed (Participants) | 9 | 9 | 9
ETDRS Letters | 54.22 (12.77) | 52.33 (16.09) | 60.22 (17.28)

4. Secondary Outcome: Best Corrected Visual Acuity (BCVA) at 28 Days After Intravitreous Dexamethasone
Description: Measure best corrected visual acuity (BCVA) at 28 days after intravitreous dexamethasone with ETDRS chart
Time Frame: 28 days after intravitreous dexamethasone
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | 0,01ml Dexamethasone Solution | 0,03 ml Dexamethasone Solution | 0,05 ml Dexamethasone Solution
Number analyzed (Participants) | 9 | 9 | 9
ETDRS letters | 58.33 (15.46) | 50.55 (18.51) | 64.11 (16.01)

5. Secondary Outcome: Intraocular Pressure (IOP) at 3 Days After Intravitreous Dexamethasone
Description: Measure intraocular pressure (IOP) 3 days after intravitreous dexamethasone - unit mmHg
Time Frame: 3 days after intravitreous dexamethasone
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0,01ml Dexamethasone Solution | 0,03 ml Dexamethasone Solution | 0,05 ml Dexamethasone Solution
Number analyzed (Participants) | 9 | 9 | 9
mmHg | 12.33 (3.90) | 13.11 (2.42) | 12.44 (3.97)

6. Secondary Outcome: Intraocular Pressure (IOP) at 28 Days After Intravitreous Dexamethasone
Description: Measure intraocular pressure (IOP) 28 days intravitreous dexamethasone - unit mmHg
Time Frame: 28 days after intravitreous dexamethasone
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0,01ml Dexamethasone Solution | 0,03 ml Dexamethasone Solution | 0,05 ml Dexamethasone Solution
Number analyzed (Participants) | 9 | 9 | 9
mmHg | 12.33 (3.16) | 12.44 (2.74) | 11.88 (2.80)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the study period - 28 days.
Description: Dexamethasone solution 4mg/ml used in the study does not have impact in cardiovascular events.
Arm/Group | 0,01ml Dexamethasone Solution | 0,03 ml Dexamethasone Solution | 0,05 ml Dexamethasone Solution
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0,01ml Dexamethasone Solution (N=9) | 0,03 ml Dexamethasone Solution (N=9) | 0,05 ml Dexamethasone Solution (N=9)
Endophthalmitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) — Incidence of endophthalmitis after intravitreous dexamethasone solution
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) — Incidence of retinal detachment after intravitreous dexamethasone solution
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0,01ml Dexamethasone Solution (N=9) | 0,03 ml Dexamethasone Solution (N=9) | 0,05 ml Dexamethasone Solution (N=9)
Intraocular pressure elevation (IOP) > 5 mmHg from baseline (Eye disorders) | 0 (0) | 0 (0) | 0 (0) — Intraocular pressure elevation > 5 mmHg from baseline or that required anti hypertensive ocular medication

LIMITATIONS AND CAVEATS:
The primary limitation of this study was the small number of participants, likely due to the strict inclusion criteria selected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT03608839/Prot_SAP_000.pdf